CLINICAL TRIAL: NCT02693899
Title: Monocentric, Biological, Uncontrolled, Prospective Study on the Feasibility of Plasma FLT3 Ligand Assay to Achieve a First Estimate of Its Prognostic Value on the Outcome of Patients Treated With Intensively for Acute Leukemia
Brief Title: Prospective Study on the Feasibility of Plasma FLT3-Ligand Assay to Achieve a First Estimate of Its Prognostic Value on the Outcome of Patients Treated Intensively for Acute Leukemia
Acronym: FLAM/FLAL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Centre de Recherche en cancérologie Nantes-Angers - CRCNA (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC15_0374
Record Dates: First submitted 2016-02-17; First posted 2016-02-29 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma (15 maximum plasma tubes of 9 mL per patient during follow-up)
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non Interventional study — The samples of the study were made in conjunction with blood tests done routinely, no additional venipuncture is provided by the study. Flt3L plasma concentration will be measured at different time monitoring of patients according to their pathology (Acute lymphoblastic leukemia or acute myeloid leukemia). The exact number of samples will vary for each patient depending on the course of the illness, it is expected up to 15 blood tubes 9mL.

SUMMARY:
Despite advances in their classification and treatment, acute leukemia remain incurable disease for the majority of patients. It is necessary to identify new prognostic markers of survival and new therapeutic targets to improve prognosis. Some studies have shown that Fms-like tyrosine kinase 3-ligand (FLT3-L) could be interesting from this. A more recent study from our group testing a novel therapy in acute lymphoblastic leukemia, showed an increase of this marker in the blood of patients responding to treatment. The aim of our prospective, non-interventional study is to measure the plasma levels of FLT3-L at different times of the management of patients with acute lymphoblastic leukemia but also myeloid. For this, analyzes of the samples collected in the usual care will be conducted to study the relationship between the plasma concentration of FLT3-L and outcomes. If there is any link, the FLT3-L could serve as a predictor of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Acute myelogenous leukemia diagnosis or lymphoblastic
* Patient intensively treated
* Patients who agreed to participate in the study and having signed the consent biocollection

Non-Inclusion Criteria:

* Patient aged under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults supported in the Clinical Hematology of the Nantes University Hospital between the beginning of the study and the end of 2017, for the diagnosis and treatment of myelogenous leukemia or acute lymphoblastic requiring intensive chemotherapy and possibly allogeneic haematopoietic stem cells.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-12-11 (Actual)

PRIMARY OUTCOMES:
Dosage of plasma FLT3-L in adult patients with acute leukemia | up to three months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PETERLIN, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No